CLINICAL TRIAL: NCT04298671
Title: Yoga-Pilates Exercise & the Effects on Urethral Rhabdosphincter Morphology and Stress Urinary Incontinence
Acronym: Y-PEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sara Cichowski, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020675
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Yoga; Pilates; Rhabdosphincter
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Pre/Post
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga-Pilates Group (Experimental): The 30-minute web-based video exercise program will combine the best yoga-Pilates exercises focused on the pelvic floor, based on prior research and expert opinion, in collaboration with yoga-Pilates instructors that participants will complete 4 times per week for 8 weeks.
  Interventions: Behavioral: Yoga-Pilates

INTERVENTIONS:
Behavioral: Yoga-Pilates — As above

SUMMARY:
This is a prospective interventional study conducted at Oregon Health & Science University that will measure the pre- and post-intervention characteristics of women with stress urinary incontinence undergoing an 8-week home yoga-Pilates intervention. The investigators plan to deliver this method of exercise to patients through a web-based video in order to increase accessibility and compliance and decrease patient costs. The investigators will assess changes using a pre- and post-treatment 1-day voiding diary, answers to questionnaires International Consultation on Incontinence Questionnaire-Short Form and Patient Global Impression of Improvement questionnaire), transperineal ultrasound, and physical exam.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) affects up to 1/3 of women and negatively impacts multiple aspects of a woman's life. Pelvic floor physical therapy has been shown to improve stress incontinence through multiple mechanisms, including rhabdosphincter hypertrophy. Yoga and Pilates have also been shown to improve stress incontinence but there is a key gap in understanding how yoga-Pilates impacts urethral function and if these exercises represent a viable option for treating SUI.

To fill this gap a new exercise is proposed: a web-based 8-week yoga-Pilates pelvic floor workout. The investigators plan to enroll women with SUI and compare urethral rhabdosphincter cross-sectional area in a pre-post intervention study. The investigators will also administer validated quality of life and severity measures for SUI to evaluate the potential efficacy of yoga-Pilates. The overarching goal of this project is to determine how yoga-Pilates impact urethral function and if these exercises decrease SUI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* >50% episodes of leakage are stress over urge incontinence on a 1-day voiding diary and/OR an answer of "when you are performing some physical activities, such as coughing, sneezing, lifting, or exercise" on the 3-Incontinence Questions (3IQ) Questionnaire
* Access to the Internet and active email address

Exclusion Criteria:

* Inability to perform yoga or Pilates due to mobility issues (specifically, inability to get up from chair without assistance or to get up from prone position on floor without assistance)
* Chronic back or neck injury that would prevent yoga or Pilates
* Dementia
* Multiple sclerosis and other neurological disorders such as stroke
* Engaged in yoga, Pilates, or pelvic floor physical therapy in past 6 months
* Current pregnancy or pregnancy in the last 6 months
* Untreated urinary tract infection (UTI), unevaluated hematuria, history of >3 diagnosed UTIs in past year
* History of bladder or rectal fistula
* Pelvic cancer or radiation
* Interstitial cystitis or chronic pelvic pain
* Congenital defect leading to urinary incontinence
* Prior anti-incontinence or urethral surgery, prior surgery for pelvic floor disorder
* Current symptomatic pelvic organ prolapse (Stage 2 or greater on exam, i.e. prolapse more than 1cm beyond the hymen)
* Majority of incontinence episodes related to urgency urinary incontinence

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Assess the change in stress urinary incontinence severity and quality of life symptoms pre/post intervention. | 8 weeks
  The investigators hypothesize that participants will report a minimally important change score difference of -2.5 utilizing the International Consultation on Incontinence Questionnaire-Short Form (range 0-21, lower scores indicate less bother from incontinence).
Estimate the effect of an 8-week intervention on urethral rhabdosphincter morphology as measured by transperineal ultrasound. | 8 weeks
  The investigators hypothesize that this program will cause hypertrophy of the urethral rhabdosphincter with an increase in urethral cross sectional area of 0.25cm2 +/- 0.6cm2.

SECONDARY OUTCOMES:
Assess the change in Patient Global Impression of Improvement (PGI-I) post-intervention | 8 weeks
  The investigators hypothesize that the majority of patients will report an answer of at least "a little better" on the PGI-I post-intervention (range 1-7; 1: "very much better", 2: "much better", 3: "a little better", 4: "no change", 5: "a little worse", 6: "much worse", 7: "very much worse")
Assess the change in number of incontinence episodes within a 24-hour period post-intervention using a 24-hour voiding diary. | 8 weeks
  The investigators hypothesize that the intervention will cause a change in number of incontinence episodes on a 24-hour voiding diary.
Assess the effect of the intervention on the levator hiatus area and anteroposterior diameter using transperineal ultrasound. | 8 weeks
  The investigators also hypothesize that the levator hiatus area and anteroposterior diameter will change over time due to hypertrophy of the levator muscles.
Assess the effect of the intervention on the degree of bladder neck descent using transperineal ultrasound. | 8 weeks
  The investigators hypothesize that the degree of bladder neck descent will change over time with Valsalva.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cichowski, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No